CLINICAL TRIAL: NCT06373042
Title: Efficacy and Safety of Tirofiban Versus Placebo After Successful Reperfusion With Endovascular Thrombectomy in Acute Ischemic Stroke Patients With Anterior Circulation Large Vessel Occlusion: a Multicenter, Double-Blind, Randomized Clinical Trial
Brief Title: Tirofiban for Successful Endovascular Stroke Thrombectomy
Acronym: ADJUVANT-2
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zhongming Qiu (Other)
Collaborators: Mianyang Central Hospital (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); The Second Hospital of Jiaozuo (Unknown); Chongzhou People's Hospital (Unknown); Xihua People's Hospital (Unknown); Xingguo People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Organization: Xinqiao Hospital of Chongqing (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADJUVANT-2
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Stroke, Acute Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Infusions, Intra-Arterial; Tirofiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban (Experimental): Intraarterial and intravenous tirofiban
  Interventions: Drug: Intraarterial and intravenous tirofiban
- Placebo (Placebo Comparator): Intraarterial and intravenous placebo
  Interventions: Drug: Intraarterial and intravenous placebo

INTERVENTIONS:
Drug: Intraarterial and intravenous tirofiban — Intraarterial and intravenous tirofiban after endovascular thrombectomy
  Other Names: Tirofiban
  Arms: Tirofiban
Drug: Intraarterial and intravenous placebo — Intraarterial and intravenous placebo after endovascular thrombectomy
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Up to 50% of acute ischemic stroke patients with large vessel occlusion failed to achieve functional independence even after successful reperfusion therapy, a phenomenon that is referred to as "futile recanalization". The mechanism of futile recanalization is complex, and some studies have shown that it may be related to factors such as tissue no reflow, reocclusion, poor status of collateral circulation, hemorrhagic transformation, impaired cerebrovascular autonomic regulation, and low perfusion volume. Several studies suggested that maximizing the improvement of cerebral reperfusion is still the primary goal of acute large vessel occlusive stroke. Structural and functional alterations in the microvascular system may be a major obstacle to reperfusion. In animal models of cerebral ischemia, downstream microvascular thrombosis may occur in the early stage of cerebral ischemia and before vascular recanalization, which is the main factor leading to incomplete reperfusion and affecting the efficacy of endovascular thrombectomy.

Mechanical thrombectomy mainly addressed the occluded large arteries, and does not consider the distal arteries. However, the recanalization of occluded large arteries does not necessarily translate into successful reperfusion of the ischemic tissue supplied by the distal capillaries. Even with complete recanalization, impaired microcirculatory reperfusion may lead to poor clinical outcomes. Therefore, we speculate that at the end of endovascular thrombectomy, microthrombi remain present in the microcirculation of brain tissue in patients with complete or near-complete cerebral angiography, and that microthrombi is more likely to be dissolved than thrombus more proximal to the heart. Therefore, intra-arterial administration of pharmaceutical, such as tirofiban, may be the only possible option to ensure complete reperfusion of ischemic tissue. Tirofiban is a platelet glycoprotein IIb/IIIa receptor antagonist, which has been widely used in acute coronary syndrome, and its role in acute ischemic stroke has attracted more and more attention from stroke experts. Previous studies have suggested that tirofiban can further increase the incidence of successful recanalization, while reducing the reocclusion rate.

Whether early administration of intraarterial and intravenous tirofiban can further improve the clinical outcomes of patients with large vessel occlusive stroke after successful mechanical thrombectomy remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Clinical inclusion criteria

  1. Aged 18 years or older;
  2. Acute ischemic stroke within 24 hours from last known well to randomization;
  3. NIHSS score ≥6 and <30 points at baseline;
  4. Written informed consent is obtained from patients and/or their legal representatives.
* Imaging inclusion criteria

  1. CTA/MRA/DSA showed occlusion of the internal carotid artery, middle cerebral artery M1 or M2 segment;
  2. For patients within 6 hours from last known well to randomization, ASPECTS 3-10 or infarct volume ≤100ml; 6-24 hours, ASPECTS 6-10 or infarct volume ≤70ml or DWI-FLAIR mismatch;
  3. Treated with endovascular thrombectomy and achieved successful reperfusion (defined as eTICI grade 2b50 or higher).

Exclusion Criteria:

1. Cardiogenic embolism;
2. Patient receive tirofiban for angioplasty/stenting prior to randomization;
3. Intracranial hemorrhage confirmed by flat panel CT on angiography machine prior to randomization;
4. Patients who are on prior anticoagulant therapy, e.g. for deep venous thrombosis or pulmonary embolism or mechanical heart valve;
5. Routine blood test platelet count less than 100×10⁹/L;
6. Renal insufficiency, glomerular filtration rate < 60 mL/min;
7. Pregnant or lactating women;
8. Allergy to tirofiban, contrast agent, nickel, titanium or its alloys;
9. History of neurological or psychiatric illness that precludes the assessment of neurological function;
10. History of bleeding disorder, severe heart, liver or kidney disease, or sepsis;
11. Any terminal illness with life expectancy less than 6 months;
12. Participating in other treatment clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Functional independence | 90 days post-randomization
  modified Rankin scale score of 0 to 2. (The modified Rankin scale scores range from 0 to 6, with 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)

SECONDARY OUTCOMES:
Recanalization on follow-up CTA or MRA | within 48 hours post-randomization
  Measured with the arterial occlusive lesion (AOL) scale
Early neurologic improvement | within 48 hours post-randomization
  defined as NIHSS score at 48 hours after randomization is reduced by 8 or more compared to NIHSS score at randomization; or the NIHSS at 48 hours after randomization is 0 to 1
Level of disability | 90 days post-randomization
  Measured with the mRS
Excellent outcome | 90 days post-randomization
  defined as mRS score of 0-1
Independent ambulation | 90 days post-randomization
  defined as mRS score of 0-3
Health-related quality of life | 90 days post-randomization
  European Quality Five-Dimension Five-Level (EQ-5D-5L) scale score
Long-term of disability level | 1 year post-randomization
  Measured with the mRS
Health-related quality of life (long-term) | 1 year post-randomization
  European Quality Five-Dimension Five-Level (EQ-5D-5L) scale score
Incidence of symptomatic intracranial hemorrhage (SICH) | within 48 hours post-randomization
  using Heidelberg criteria to assess SICH
Radiologic intracranial hemorrhage rate | within 48 hours post-randomization
  using Heidelberg criteria to assess SICH
Mortality | 90 days post-randomization
  Death from any cause
Incidence of non-hemorrhagic serious adverse events | 90 days post-randomization
  such as pneumonia, respiratory failure, circulatory failure, cerebral herniation, secondary epilepsy, sepsis, renal failure, acute coronary syndrome, venous thrombosis, etc

CONTACTS AND LOCATIONS:
Overall Officials: Zhongming Qiu, MD, Principal Investigator — The 903rd Hospital of PLA, China

IPD SHARING:
Plan to Share IPD: Yes
study data without patient information
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Related papers published 3 months later, the IPD will be shared.
Access Criteria: qiuzhongmingdoctor@163.com